CLINICAL TRIAL: NCT06004271
Title: The Effect of Kinesio Taping on q Angle and Pes Planus in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar68
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy; Pes Planus
Keywords: Cerebral palsy; Kinesio tape; Pes Planus; Q angle; Exercise
MeSH Terms: conditions — Cerebral Palsy; Flatfoot; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomization will be made and divided into 3 groups with equal number of participants. The groups will be called control, experiment, and placebo. Only physiotherapy will be applied to the control group, kinesio taping and physiotherapy to the experimental group, and damask taping and physiotherapy to the placebo group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): In the control group, only the exercise program was applied and the first and last measurements will be compared.
  Interventions: Other: exercise
- experimental group (Experimental): In the experimental group, kinesiology taping will be applied twice a week for 8 weeks together with exercise. Kinesiology taping was first applied by closing the malleoli from the upper part of the foot, and stretching it to the anterior capsule of the foot using the ligament technique. For the second tape, it covered the plantar area under the malleolus and was attached in the form of stirrups. During the application, the tape will be applied with full tension on the malleolus and 50-75% tension will be applied on the other parts.
  Interventions: Other: exercise; Other: exercise and taping
- placebo group (Placebo Comparator): Tape application will be applied in the placebo group as it was in the experimental group. Kinesiology taping will be attached horizontally without tension along the Tensor Facie Late line. The application to the ankle will be attached horizontally without tension slightly above the lateral malleolus.
  Interventions: Other: exercise; Other: placebo

INTERVENTIONS:
Other: exercise — Exercise protocol:
  Progressive Resistance Exercise Training Bridge exercise sit-up exercise functional walking exercise Stretching
Other: exercise and taping — When applying kinesiology taping to the gluteus medius, first of all, for its anterior fiber, the tape portion will be attached lateral to the Spina iliaca anterior superior by giving a slight slope downwards from the crista iliaca with 50-75% tension. For the posterior fiber; Starting from the trochanter major, 50-75% tension will be applied along the muscle fiber.
  Arms: experimental group
Other: placebo — In the placebo tape application, the kinesiological tappings will be adhered horizontally without tension along the long line of the Tensor facie late muscle. The application to the ankle will be attached horizontally, without tension, slightly above the lateral malleolus.
  Arms: placebo group

SUMMARY:
The aim of our study is to examine the effect of using kinesiology tape and using it for 8 weeks on Q angle and pes planus on children with cerebral palsy.

DETAILED DESCRIPTION:
At the beginning of the study, the pes planus level of the children will be determined. Then randomization will be made and divided into 3 groups with equal number of participants. The groups will be called control, experiment, and placebo. Only physiotherapy will be applied to the control group, kinesio taping and physiotherapy to the experimental group, and damask taping and physiotherapy to the placebo group. The study will be followed for 8 weeks, and pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with cerebral palsy
* Gross Motor Function Classification System level 1,2 and 3
* 2-18 years

Exclusion Criteria:

* Having Gross Motor Function Classification System levels 4 and 5
* Those with genetic and metabolic diagnosis

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Calcaneo-tibial angle measurement | 10 weeks
  The calcaneo-tibial angle measurement is a method used in the general evaluation of the foot. By measuring this angle, it is checked whether the problems in the foot are related to the rear foot. Normal values in this measurement are eversion angles between 4° and 8°. During the evaluation, the angle between the axis passing through the middle of the calcaneus and the place where the Achilles tendon attaches to the calcaneus will be measured, while the patient is in the prone position, not putting weight on his foot. Measurements will be made again while standing on the ground. Each measurement will be repeated 3 times. The differences between the results obtained during standing and prone lying will be calculated. The measurements will be averaged and recorded.
Navicular bone drop test | 10 weeks
  This assessment method evaluates midfoot mobility and medial longitudinal arch depression. In this method, the measurements should be between 5-9 mm. Before the evaluation, the height of the tubercle of the navicular bone will be measured in meters in millimeters, while the patient is in a sitting position, not putting weight on his feet. Then, the patient will be lifted up, and the patient will be asked to give equal weight to both feet in an upright position, and the measurement will be repeated 3 times. The average of the measurements will be recorded after they are taken. After the measurement, the difference between standing and in bed will be found.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan SANCAKDAR, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Üsküdar, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Armstrong RW. Definition and classification of cerebral palsy. Dev Med Child Neurol. 2007 Mar;49(3):166. doi: 10.1111/j.1469-8749.2007.00166.x. No abstract available. PMID 17355470
- [Background] Shakeri H, Keshavarz R, Arab AM, Ebrahimi I. Clinical effectiveness of kinesiological taping on pain and pain-free shoulder range of motion in patients with shoulder impingement syndrome: a randomized, double blinded, placebo-controlled trial. Int J Sports Phys Ther. 2013 Dec;8(6):800-10. PMID 24377066
- [Background] Shultz SJ, Nguyen AD, Windley TC, Kulas AS, Botic TL, Beynnon BD. Intratester and intertester reliability of clinical measures of lower extremity anatomic characteristics: implications for multicenter studies. Clin J Sport Med. 2006 Mar;16(2):155-61. doi: 10.1097/00042752-200603000-00012. PMID 16603886
- [Background] Park EY, Kim WH. Structural equation modeling of motor impairment, gross motor function, and the functional outcome in children with cerebral palsy. Res Dev Disabil. 2013 May;34(5):1731-9. doi: 10.1016/j.ridd.2013.02.003. Epub 2013 Mar 15. PMID 23500167
- [Background] Merino-Andres J, Garcia de Mateos-Lopez A, Damiano DL, Sanchez-Sierra A. Effect of muscle strength training in children and adolescents with spastic cerebral palsy: A systematic review and meta-analysis. Clin Rehabil. 2022 Jan;36(1):4-14. doi: 10.1177/02692155211040199. Epub 2021 Aug 18. PMID 34407619